CLINICAL TRIAL: NCT05807269
Title: Prevention and Rehabilitation of Stroke in Uganda
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Gunilla Eriksson, Principal investigator, Karolinska Institutet
Other Study IDs: 2022-04303
Record Dates: First submitted 2023-03-13; First posted 2023-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with stroke: Participants with stroke or risk factors for stroke

SUMMARY:
Stroke is increasing in low-income countries in Africa, and knowledge is lacking on risk factors and how to prevent stroke as well as how to best use the resources for rehabilitation after stroke which are very limited. Knowledge generation within this area is therefore urgently needed. This collaboration between the research group HELD (Health and Everyday Life among people with neurological Disorders), Karolinska Institutet (KI) and the research surveillant site Africa Medical and Behavioral Sciences Organization (AMBSO) population health surveillance (PHS), will create substantial research opportunities to develop and improve prevention and rehabilitation for stroke, which is in line with the sustainable development goals to reduce the prevalence and mortality rates due to NCDs. AMBSO is collecting data from 17 000 households on many potential risk factors for stroke. Questions about stroke primary and secondary prevention of stroke and impact of stroke or need of rehabilitation could be added to the existing questionnaires such as the validated Ugandan version of the Stroke Impact Scale. This is intended to fulfill the aim of the network which is to increase the knowledge of occurrence and consequences of NCDs with a specific focus on stroke, which will be valuable for the development of preventive healthcare policy documents and guidelines for appropriate prevention strategies and rehabilitation interventions.

Research questions in relation to NCDs with focus on stroke prevention and rehabilitation:

* How many cases (prevalence) are reported in the targeted study sites and what is the mortality rate (incidence) that can specifically relate to stroke?
* How does stroke and other NCDs affect and impact the quality of life for persons living in Uganda?
* Which factors impact the recovery process after stroke?
* What sort of rehabilitation is needed in the study areas for persons affected by stroke? In addition, risk factors of stroke such as diabetes and hypertension will be mapped.

ELIGIBILITY:
Inclusion Criteria:

* Stroke
* Risk factors for stroke: hypertension, diabetes, HIV, malaria, physical inactivity, obesity

Exclusion Criteria:

* Not having had stroke and/or having no risk factor for stroke

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample from Wasiko and Hoima in Uganda
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Stroke Impact Scale-16 | At one assessment point during 2023-2024
  Questionnaire comprising 16 statements concerning perceived impact of stroke. Each item is rated on a scale from 0 (high impact) to 5 (no impact).
Stroke Impact Scale, perceived recovery | At one assessment point during 2023-2024
  Perceived recovery after stroke is rated on a visual analogue scale ranging from 0 (no recovery) to 100 (full recovery).

SECONDARY OUTCOMES:
Life Satisfaction Checklist (LISat-11) | At one assessment point during 2023-2024
  Questionnaire that assesses life satisfaction with one global item "Life as a whole", and 9 domain-specific items. Answering alternatives range from 1 (very dissatisfied) to 6 (very satisfied)
Patient Health Questionnaire-9 | At one assessment point during 2023-2024
  Questionnaire with nine items that inquire about the frequency of depressed mood and anhedonia over the past two weeks. Score ranges from 0 (not at all) to 6 (nearly every day) where higher scores indicate higher frequency of depressed mood
Generalized Anxiety Disorder Assessment-7 | At one assessment point during 2023-2024
  A questionnaire assessing generalized anxiety disorder. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
Health Literacy Questionnaire | At one assessment point during 2023-2024
  Questionnaire that assesses health literacy. The Health Literacy Questionnaire contains 44 items, which are divided into nine areas of health literacy. The first five scales are scored on a 4-point Likert scale (ranging from strongly disagree to disagree, agree, and strongly agree), building part I. The other four scales, representing part II, are scored on a 5-point Likert scale where respondents are asked to rate the level of difficulty in undertaking a task (ranging from cannot do, always difficult, usually difficult, sometime difficult, usually easy, and always easy). Higher scores indicate better health literacy. In total six selected questions from part I and part II are used.
Use of health care services | At one assessment point during 2023-2024
  Six questions on use of healthcare services, and information received on stroke and its consequences.
Question about quality of life | At one assessment point during 2023-2024
  The respondents are asked to rate their quality of life on a on a five-point scale from 1 (very poor) to 5 (very good)

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Eriksson, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Uganda (2):
  - AMBSO, Hoima, Hoima
  - AMBSO, Wakiso, Kampala

IPD SHARING:
Plan to Share IPD: No